CLINICAL TRIAL: NCT04102527
Title: Evaluation of the Impact of Transit Troubles in Patients Undergoing Peritoneal
Brief Title: Evaluation of the Impact of Transit Troubles in Patients Undergoing Peritoneal Dialysis
Acronym: TransDiPe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Vichy (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHV 2018-1
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Peritoneal Dialysis Complication; Constipation
MeSH Terms: conditions — Constipation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with Terminal Chronic Kidney Disease undergoing Peritoneal Dialysis for at least three months in stable condition
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients have to complete the study questionnaires every 2 months :
  * Digestive Functional Score of Neurological Patients
  * Bowel Function Index
  * Severity score for constipation
  * Bristol Scale
  * Constipation assessment scale
  * Estimate scale of risk of constipation

SUMMARY:
Patients with Terminal Chronic Kidney Disease undergoing Peritoneal Dialysis (PD) often have pathophysiological factors that promote chronic constipation. It affects the quality of life of Patients undergoing PD in a much greater way than for hemodialysis patients because it causes complications, mechanical and infectious associated with the transmural migration of enteral bacteria, with an impact on patient morbidity and survival of the technique. In addition, it should be noted that PD patients often take potentially constipants treatments such as phosphorus chelators, calcium inhibitors, opiates, iron preparation and antidepressants. Taking these drugs decreases gastric acidity, which is associated with an increased prevalence of peritonitis.

In this context, a significant lack of literature, specifically studying the risk factors for constipation in Terminal Chronic Kidney Disease patients treated with DP and the correlation with mechanical and infectious complications, is improvable.

DETAILED DESCRIPTION:
Patients included in this trial will be monitored as part of the usual management of their pathology, a Terminal Chronic Kidney Disease treated by the Peritoneal Dialysis technique.

During this treatment, patients will be follow every 2 months in consultation in the Metabolic Diseases Department of the Hospital of Vichy.

These consultations include:

* Pre-selection consultation/Inclusion (visit to J0 -3 months)
* Half-yearly review (visit J0, visit at 12 months and visit at 24 months)
* Simple consultation (visits to 2, 4, 8, 10, 14, 16, 20, 22 months)
* Annual review (visits at 6 and 18 months)

In this prospective trial, there is no intervention on the patient; They will only have to complete questionnaires on their intestinal transit (Charlson Scale, Katz Scale, Neurological Functional Score, Intestinal Function Index, Severity Score for constipation, Bristol Scale, Constipation Assessment Scale, Constipation Risk Assessment Scale). No minimal risk and constraint is identified, excluding our trial from the category of interventional research. The category 3 (non-interventional trial) of the jardé classification is therefore accepted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TerminalChronic Kidney disease undergoing Peritoneal Dialysis for at least three months in stable condition,
* Patients who are able to complete the study questionnaires every 2 months,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Ability to understand the French language for an informed understanding of the information and non-opposition forms,
* Affiliation with the French Social Security scheme.

Exclusion Criteria:

* Patients whose peritoneal dialysis catheter is considered non-functional at J0,
* Patients with a medical and/or surgical history considered by the investigator or his representative to be not compatible with the trial,
* Patients with unstabilized progressive pathology at the time of inclusion at J0,
* Patients who are mentally incapacitated to answer questionnaires,
* Women of childbearing age who do not use an effective contraceptive method, pregnant or lactating women.
* Patients with legal protection measures (curatorship, guardianship, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable patients who have been in Peritoneal Dialysis for at least three months will be pre-selected three months before the start of the study and included via the Metabolic diseases Center of the Hospital.
  This protocol will be offered to adult patients suffering from Terminal Chronic Kidney disease undergoing Peritoneal Dialysis.
  The investigator will inform the details of the protocol and answer all questions from patients. It will be given sufficient time to reflect for the signing of the information and non-opposition form. Volunteers will be included after signing this document.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine whether there is a relationship between transit disorders and the rate of digestive germ peritonitis in patients with Terminal Chronic Kidney disease on Peritoneal Dialysis | 4 years
  The investigators will count the number of peritonitis associated with transit disorders in patients with Terminal Chronic Kidney Disease undergoing Peritoneal Dialysis

SECONDARY OUTCOMES:
To determine whether there are variations in the relationship between transit disorders and the rate of peritonitis depending on the therapeutic management of these transit disorders. | 4 years
  To assess the existence of an episode of peritonitis from all causes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital center, Vichy, France

IPD SHARING:
Plan to Share IPD: No
Source documents defined as any original document or object to prove the existence or accuracy of a data or fact recorded during the clinical study will be kept for 15 years by the Hospital Center; this is the hospital medical record, original results of the patient's biological examinations.
  The protocol data that will be collected in the observation book and which will be considered source data can be found in the attached observation book.
  Source data will be collected by the service's investigators and nurses; It will be collected in the CRF by investigators.
  The data will then be entered into the Excel database by the clinical research officer and a team member (investigator, intern or IDE) for a double entry.
  During or after the research, data collected on the appropriate individuals and transmitted to the sponsor by investigators will be anonymized.